CLINICAL TRIAL: NCT01357681
Title: Effects of EGCG (Epigallocatechin Gallate) in Huntington's Disease The ETON-Study - A Randomized, Double-blind, Stratified, Placebo-controlled Prospective Investigator Initiated Multicenter Trial -
Brief Title: Effects of EGCG (Epigallocatechin Gallate) in Huntington's Disease (ETON-Study)
Acronym: ETON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Josef Priller, Prof. Dr. med; Director, Department of Neuropsychiatry, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-023941-31
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Huntington Disease
Keywords: Huntington Disease; Cognition; Motor; Behaviour; Functional Capacity; Quality of Life; Biomarker; MRI; Huntingtin; EGCG
MeSH Terms: conditions — Huntington Disease; Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (2)-epigallocatechin-3-gallate (EGCG) (Experimental): Month 01:400 mg /day (200-0-200) p.o. Month 02:800 mg /day (400-0-400) p.o. Month 03 -12: 1200 mg /day (600-0-600) p.o.
  Interventions: Drug: (2)-epigallocatechin-3-gallate (EGCG)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: (2)-epigallocatechin-3-gallate (EGCG) — Month 01:400 mg /day (200-0-200) Month 02:800 mg /day (400-0-400) Month 03 -12: 1200 mg /day (600-0-600)
  Arms: (2)-epigallocatechin-3-gallate (EGCG)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Huntington's disease (HD) is an inherited autosomal dominant, progressive neurodegenerative disease. Clinically, HD is characterized by a triad of movement disorders, cognitive impairments and psychiatric disturbances. These symptoms represent a tremendous burden for patients and caregivers. HD is a fatal disorder with neither cure, nor evidence-based standard therapy available.

The green tea polyphenon (2)-epigallocatechin-3-gallate (EGCG) was shown to have beneficial effects in cell and animal models of HD. The aim of this study is to evaluate the efficacy and tolerability of EGCG in HD.

The investigators hypothesize that Sunphenon EGCG administered at a maximal daily dose of 1200 mg compared to placebo during a period of 12 months improves cognition in patients with HD. As primary outcome measure, the change of cognitive functions (as measured by the Unified Huntington's Disease Rating Scale (UHDRS)-Cognition composite score of Stroop test, Verbal fluency & Symbol Digit Modalities Test) after 12 months in comparison to Baseline was defined.

The investigators further expect a positive influence of EGCG on other clinical manifestations of HD, measurable effects of EGCG on HD biomarkers and good safety and tolerability of EGCG in HD patients.

ELIGIBILITY:
Inclusion Criteria:

* Chorea Huntington (CAG repeats >39)
* UHDRS TFC >5
* ≥18 years of age
* Readiness and ability to take oral medication
* Normal liver function laboratory test
* Stable concomitant medication regimen > 4 weeks prior to Baseline
* Motivation for women with childbearing potential to use highly efficient contraception

Exclusion Criteria:

* Clinically relevant abnormal findings in the ECG, vital signs, physical examination or laboratory values at Screening,
* Long-term treatment with potentially hepatoxic medication
* Any unstable medical condition
* BDI Depression score > 9 AND clinical diagnosis of depression
* Suicidal tendencies
* Cognitive dysfunction defined as a score < 23 in the Mini-Mental State Examination (MMSE) at Screening
* Liver or renal disease
* Schizophreniform psychosis within the last 6 months before baseline
* Consumption of more than two cups of black tea per day, consumption of green tea, consumption of > 500 ml /day of grapefruit juice
* Participation in other Arzneimittelgesetz (AMG) or Medizinproduktegesetz (MPG) studies (three months before and during participation)
* Pregnancy/ lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change of cognitive functions (UHDRS-Cognition: composite score of Stroop test, Verbal fluency & Symbol Digit Modalities Test) after 12 months in comparison to baseline | Month 0, Month 12

SECONDARY OUTCOMES:
UHDRS Motor Score | Month 0, Month 12
UHDRS Behavioural Score | Month 0, Month 12
UHDRS Functional Assessment | Month 0, Month 12
UHDRS Total Functional Capacity (TFC) | Screening, Month 12
Clinical Global Impression (CGI) | Month 0, Month 12
Depression: Beck Depression Inventory (BDI) | Screening, Month 1, Month 2, Month 3, Month 6, Month 9, Month12, Month 13
Health-related Quality of Life: Short Form (36) Health Survey (SF-36) | Month 0, Month 12
Subjective Well-Being: Satisfaction With Life Scale (SWLS) | Month 0, Month 12, Month 13
Affective Processing: Positive and Negative Affect Schedule (PANAS) | Month 0, Month 12, Month 13
Tonic and phasic Alertness | Month 0, Month 12
Global Cognition: Mini Mental State Examination | Screening, Month 12, Month 13
Quantitative evaluation of motor functions: Qmotor | Month 0, Month 12
Brain atrophy: assessed by magnetic resonance imaging (MRI)-voxel-based morphometry (VBM) | Month 0, Month 12
Pharmacokinetics and tolerability of EGCG | Month 1 - Month 12
  assessment of side effects and determination of blood and cerebrospinal fluid (CSF) levels of EGCG
Determination of huntingtin expression levels | Screening - Month 13
  Quantification of huntingtin in blood and CSF (optional)

CONTACTS AND LOCATIONS:
Overall Officials: Josef Priller, MD, Principal Investigator — Department of Neuropsychiatry, Charité Universitätsmedizin Berlin, Germany
Locations (3):
- Germany (3):
  - Department of Neuropsychiatry, Berlin
  - Neurologische Klinik der Ruhr-Universität Bochum, Bochum
  - Universitätsklinikum Ulm, Klinik für Neurologie, Ulm